CLINICAL TRIAL: NCT04652011
Title: Long-term Management of Patients With Benign Gynecological Pathology and Chronic Pelvic Pain and Follow-up After Minimally Invasive Surgery
Brief Title: Long-term Management of Patients Surgically Treated for Chronic Pelvic Pain by Minimally Invasive Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Carlo Alboni, MD, PhD, Dr. Carlo Alboni MD, PhD Head of Minimally Invasive and Robotic Gynecologic Surgery Unit University Hospital of Modena - Italy, Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: 0024582/19
Record Dates: First submitted 2020-11-16; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Pelvic Pain
Keywords: Pelvic Pain; Endometriosis; Minimally invasive Surgery
MeSH Terms: conditions — Pelvic Pain; Endometriosis | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic pelvic pain: Patients with chronic pelvic pain and a benign gynecologic disease associated, referring to our Unit, medically or surgically treated from 2010 to 2019
  Interventions: Procedure: Minimally Invasive Gynecologic Surgery; Procedure: osteopathic manipulative treatment; Drug: Pain killer

INTERVENTIONS:
Procedure: Minimally Invasive Gynecologic Surgery — Minimally Invasive Surgery for gynecologic disease (laparoscopy, robotic surgery, vaginal surgery)
Procedure: osteopathic manipulative treatment — Osteopathic manipulative treatment
Drug: Pain killer — Common pain killer (paracetamol, Ibuprofen, ketoprofen)

SUMMARY:
It is a retrospective observational study based on the analysis of the medical records of patients treated for chronic pelvic pain and benign gynecological pathologies at the Gynecology Unit of the University Hospital of Modena from 2010 to 2019. The aim of the study is to analyze the effects of medical and surgical treatments on chronic pelvic pain and associated pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Underwent Minimally invasive gynecologic surgery from 2010 to 2019
* Chronic pelvic pain
* Benign gynecologic disease (Endometriosis, myoma, adenomyosis, pelvic organ prolapse

Exclusion Criteria:

* malignant gynecologic disease
* chronic pelvic pain not linked to gynecologic disease

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pelvic pain and a benign gynecologic disease associated, referring to Gynecologic Unit of University Hospital of Modena, who underwent minimally invasive surgery from 2010 to 2019
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Pain Scores on the Numeric Rating Scale at 6 months after surgery | Baseline and 6 months after surgery
  Change From Baseline in Pain Scores on the Numeric Rating Scale at 6 months after surgery
Change From Baseline in Pain Scores on the Numeric Rating Scale at 6 months after Osteopathic manipulative treatment | Baseline and 6 months after Osteopathic manipulative treatment
  Change From Baseline in Pain Scores on the Numeric Rating Scale at 6 months after Osteopathic manipulative treatment

SECONDARY OUTCOMES:
Change From Baseline in constipation on the constipation score system (CSS) by Agachan-Wexner at 6 months after surgery | Baseline and 6 months after surgery
  Change From Baseline in constipation on the constipation score system (CSS) by Agachan-Wexner at 6 months after surgery
Analysis of postoperative complications using Clavien-Dindo classification | 1 month after surgery
  Analysis of postoperative (1 month after surgery) complications using Clavien-Dindo classification
Incidence of endometriosis among patients with chronic pelvic pain | Baseline
  Incidence of endometriosis among patients with chronic pelvic pain

CONTACTS AND LOCATIONS:
Locations (1):
- Carlo Alboni, Modena, Italy

IPD SHARING:
Plan to Share IPD: No
I prefer to not share individual participant data